CLINICAL TRIAL: NCT01056029
Title: An Open Label, Single-Arm, Dose-Escalation Phase 1 Study of G-202 (Mipsagargin) in Patients With Advanced Solid Tumors
Brief Title: Dose-Escalation Phase 1 Study of G-202 (Mipsagargin) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GenSpera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G-202-001
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Advanced Solid Tumors
Keywords: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- G-202 (Experimental)
  Interventions: Drug: G-202

INTERVENTIONS:
Drug: G-202 — Thapsigargin is Pro-drug chemotherapy which will be administered by intravenous infusion over 1 hour on Days, 1, 2 and 3 of each 28 day cycle

SUMMARY:
This is an open-label, single-arm, dose-escalation Phase I study to determine the maximum tolerated dose (MTD) of G-202 (mipsagargin) when administered once daily for 3 consecutive days of a 28-day cycle in patients with advanced solid tumors. G-202 will be administered by intravenous infusion over 1 hour on Days 1, 2 and 3 of each 28-day cycle.

DETAILED DESCRIPTION:
Pro-drug chemotherapy is an approach to cancer treatment that is being investigated as a means to achieve higher concentrations of cytotoxic or biologically active agents at a tumor location while avoiding systemic toxicity. With pro-drug chemotherapy, a relatively non-toxic form of a cytotoxin, the pro-drug, is converted into the active cytotoxic agent at the tumor site or other specific location. G-202 (mipsagargin) is a thapsigargin pro-drug; it consists of a cytotoxic analog of thapsigargin coupled to a masking peptide which inhibits its biologic activity until proteolytic cleavage at the tumor site. Thapsigargin is a natural product with profound effects on cell viability. Thapsigargin is a non-cell-type specific toxin with documented ability to kill a broad spectrum of cancer cell lines as well as normal endothelial cells, fibroblasts and osteoblasts. It induces a rapid and pronounced increase in the concentration of cytosolic calcium, due to blockade of the Sarcoplasmic/Endoplasmic Reticulum Calcium ATPase (SERCA) pump to which it binds with high affinity. The increase in cytosolic calcium leads to induction of apoptosis and ensuing cell death.

The anti-tumor effect of G-202 in humans with advanced solid tumors is not yet known.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed malignancy that is metastatic or unresectable and for which standard curative measures do not exist or are no longer effective
* Disease that is measurable and/ or evaluable by RECIST criteria. Patients with prostate cancer require presence of disease on bone scan and/or CT scan and evidence of increasing PSA after standard hormonal therapy
* ECOG Performance Status ≤ 2
* Life expectancy estimated to be at least 3 months
* Acceptable liver function:

  * In the absence of disease involvement in the liver and if bilirubin ≤ 1.5 times institutional upper limit of normal (ULN), AST (SGOT), ALT (SGPT) and GGT may be ≤ 2 times ULN
  * In the presence of disease involvement in the liver and if bilirubin ≤ 1.5 times institutional upper limit of normal (ULN), AST (SGOT), ALT (SGPT) and GGT may be ≤ 5 times ULN
  * Alkaline phosphatase ≤ 2.5 times ULN Patients with bone metastases alkaline phosphatases ≤ 5 times ULN
* Acceptable renal function:

  * Serum creatinine ≤ 1.5 times ULN, OR
  * Calculated creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula)
* Acceptable hematologic status:

  * Absolute neutrophil count (ANC) ≥ 1500 cells/mm3 (1.5 ×109/L)
  * Platelet count ≥ 100,000 platelet/mm3 (100 ×109/L)
  * Hemoglobin ≥ 9 g/dL
* Urinalysis with no evidence of proteinuria
* Acceptable coagulation profile (PT or INR, PTT) < 1.5 times ULN
* At least 4 weeks since prior chemotherapy or surgery, with recovery to Grade 1 or baseline of significant toxicities felt related to prior drug(s)
* Women of childbearing potential must have a negative serum pregnancy test at screening.
* All patients (males and females) of child-bearing potential must agree to use an effective method of birth control
* Ability to understand and willingness to sign a written informed consent document
* Patients with prostate cancer must continue androgen deprivation therapy with LHRH agonists

Exclusion Criteria:

* Documentation of keratosis follicularis, also known as Darier or Darier-White disease
* Known hypersensitivity to any study drug component, including thapsigargin derivatives, Polysorbate 20, or propylene glycol
* Patients with known and untreated brain metastases. Patients with brain metastases that have been treated and demonstrated to be clinically stable for at least 30 days may be enrolled onto the study
* Patients with a family history of coagulopathy or patients with DVT or pulmonary embolus within the last 6 months
* Patients taking anti-coagulants that include Coumadin or low molecular weight heparin
* Patients with pre-existing cardiac conditions:

  * Prior documented myocardial infarction within the last 6 months
  * Pre-existing cardiac failure (NYHA class III-IV)
  * Atrial fibrillation on anti-coagulants
  * Unstable angina
  * Severe valvulopathy
  * Cardiac angioplasty or stenting within the last 6 months
* Use or requirement for use of inhibitors or inducers of cytochrome isoenzymes
* Corrected QTc prolongation value, calculated using Bazett's formula (QTcB = QT/RR ½), > 450 msec
* Pregnant or lactating females
* Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study
* Active uncontrolled infection, including known history of AIDS or hepatitis B or C
* Any psychological, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule
* Concurrently receiving any other investigational agents while on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Determine the MTD and DLT(s) of G-202 administered by intravenous infusion daily for 3 consecutive days on a 28-day cycle in patients with advanced solid tumors. | 2 years
Establish the recommended dose of G-202 to be used in Phase II studies. | 2 years
Determine the pharmacokinetics of G-202 administered by intravenous infusion daily for 3 consecutive days on a 28-day cycle in patients with advanced solid tumors. | 2 years

SECONDARY OUTCOMES:
Investigate the safety profile of G-202 administered by intravenous infusion daily for 3 consecutive days on a 28-day cycle in patients with advanced solid tumors. | 2 years
Document any evidence of anti-tumor activity, including response rate, disease stability, progression-free or overall survival, in response to G-202 administration | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: George Wilding, M.D, Principal Investigator — University of Wisconsin, Madison; Michael Carducci, M.D., Principal Investigator — Johns Hopkins University; Devalingam Mahalingam, MD, Principal Investigator — University of Texas, Health Science Center,Cancer Therapy and Research Center
Locations (3):
- United States (3):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - University of Texas, Health Science Center,Cancer Therapy and Research Center, San Antonio, Texas
  - University of Wisconsin Paul P Carbone Comprehensive Cancer Center, Madison, Wisconsin